CLINICAL TRIAL: NCT05275738
Title: The Glaucoma Nicotinamide Trial - A Prospective, Randomized, Placebo-controlled, Double-masked Trial
Brief Title: The Glaucoma Nicotinamide Trial
Acronym: TGNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Center for Eye Research Australia (Other); Karolinska Institutet (Other); Singapore National Eye Centre (Other Government); Duke-NUS Graduate Medical School (Other); University of Melbourne (Other); University of Adelaide (Other); Lund University (Other); Linkoeping University (Other Government); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGNT; SGNT (Other: Umeå University); VBIGS (Other: Centre for Eye Research Australia)
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Glaucoma
Keywords: Neuroprotection; Glaucoma; Nicotinamide
MeSH Terms: conditions — Glaucoma | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both patients, care givers and investigators are masked to the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Active Comparator): Participants will receive 750mg nicotinamide tablets 1+1 per day (1.5g) for 6 weeks and after that 2+2 per day (3.0g).
  Interventions: Dietary Supplement: Nicotinamide
- Placebo (Placebo Comparator): Participants will receive 750mg placebo tablets 1+1 per day for 6 weeks and after that 2+2 per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide — Study tablets for nicotinamide are produced by Blackmores Ltd.
  Arms: Nicotinamide
Other: Placebo — Study tablets for placebo are produced by Blackmores Ltd.
  Arms: Placebo

SUMMARY:
The Glaucoma Nicotinamide Trial (TGNT) is a prospective, randomized, placebo-controlled double-masked clinical trial composed of two cohorts; The Swedish Glaucoma Nicotinamide Trial (SGNT) and the Vitamin B3 In Glaucoma Study (VBIGS). Patients with open-angle glaucoma (OAG) will be randomized to receive either Nicotinamide or placebo through block randomization stratified by glaucoma subtype with a 1:1 allocation.

DETAILED DESCRIPTION:
The treatment arms that included patients will be randomized into are either Nicotinamide tablets 1.5g for 6 weeks and then 3.0g onwards or true placebo tablets. A major difference between the SGNT and VBIGS is that in SGNT untreated newly diagnosed glaucoma patients will be included whereas in VBIGS glaucoma patients with intraocular pressure lowering treatment will be included. Also, in SGNT an additional non-blinded arm with healthy subjects will receive Nicotinamide tablets 1.5g for 6 weeks and then 3.0g onwards. For participants where both eyes are eligible, both will be included.

The primary endpoint is visual field progression change over two years.

ELIGIBILITY:
SGNT:

Inclusion Criteria:

* Adult participants (>18 years) with newly-diagnosed and previously untreated POAG or PEXG in one or both eyes. Glaucoma is defined as reproducible visual field (VF) defects that cannot be explained by other disease or damage, and a suspect/abnormal optic nerve head and/or nerve fibre layer defect.
* Participants need to have visual acuity of Snellen ≥ 6/12 (0.5) or better.
* Have performed at least two reliable VFs (SITA-Fast 24-2), with <33% fixation losses and <15% false positives

Exclusion Criteria:

* VF damage worse than -10dB in the best eye and -16dB in the worse eye or a paracentral spot with -10dB or less in any eye),
* IOP >35mmHg in any eye or a mean IOP of 30mmHg or higher (two measurements), •inability to perform VFs,
* pregnancy/breastfeeding,
* those unwilling to abstain from NAM supplements,
* allergic to NAM/niacin,
* diagnosed with cancer in the last 5 years (except treated basal or squamous cell carcinoma),
* a history of liver disease or stomach ulcers,
* disease that prevents long-term follow-up,
* neurologic or other non-glaucomatous conditions apart from cataract that may affect the VF, •inability to understand and speak Swedish or English,
* a history of intraocular surgery (apart from uncomplicated cataract surgery) and
* diseases that are known to affect retinal function (e.g. > mild age-related macular degeneration, > stage I diabetic retinopathy).

VBIGS:

Inclusion Criteria:

* Patients aged 18 years or older, with definitive, treated POAG including normal tension glaucoma, PEXG in both eyes
* Best-corrected visual acuity ≥ 6/18
* Severity of visual field loss, MD between -3 and -18 dB. This range includes people with moderate disease which optimises detection of progression.
* Patient must have performed at least two reliable VFs (24-2), with <33% fixation losses and <15% false positives.
* Previous selective laser trabeculoplasty is acceptable (IOP-lowering laser treatment) if 3 or more months prior, and normal liver function tests.
* Those taking NAM already will undergo a 1-month washout period before commencing the study.

Exclusion Criteria:

* Patients with a history of hepatic disease, gout, visually significant cataracts, other conditions that can affect VF results, cataract surgery in the last 3 months or glaucoma filtration surgery in last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual field progression | Two years
  Change in rate of progression between the two study arms

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - S:t Eriks Eye Hospital, Stockholm
  - Umeå University, Umeå